CLINICAL TRIAL: NCT02090270
Title: Hair Cortisol and the Risk of Stroke
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC-13-0275-CTIL
Record Dates: First submitted 2014-03-12; First posted 2014-03-18 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2015-01

CONDITIONS: ISCHEMIC STROKE
Keywords: hair cortisol; stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ischemic stroke: Sudden onset of focal neurologic deficit lasting more than 24 hours, with cerebral hemorrhage ruled out by brain CT, in the absence of obvious causes of embolic stroke.
- Control: Patients admitted to an internal medicine department for indications other than stroke or acute myocardial ischemia.

SUMMARY:
The purpose of this study is to prospectively examine the relation between ischemic stroke and hair cortisol concentration. The investigators hypothesize that patients with ischemic stroke have higher levels of hair cortisol compared to controls.

DETAILED DESCRIPTION:
Acute physical and emotional stressors are well known triggers of cardiovascular events. However, it is not clear whether the same association exists with chronic stress. Data on this issue have been limited by lack of adequate clinical studies and inconclusive results. One of the possible explanations may be the absence of a reliable mode for quantitative assessment of chronic stress. To date, studies on the effects of chronic stress on cardiovascular events have used psychosocial questionnaires. These are subject to recall bias, as having an event may stimulate the patient to strive harder to identify previous stressors. Furthermore, most studies on the association of chronic stress and cardiovascular events have focused on acute coronary events, and only few have examined the association with stroke.

Both physical and emotional stress activate several neuroendocrine systems, the most important being the hypothalamic-pituitary-adrenal (HPA) axis that stimulates the production and secretion of glucocorticoids (especially cortisol) from the adrenal cortex. Therefore, cortisol is considered to be a "stress hormone" and higher levels of serum cortisol have been observed in patients with acute stress such as those presenting with acute myocardial infarction and stroke compared to healthy controls. Moreover, it has been shown that serum cortisol levels correlates with the severity of the disease and adverse outcome in patients presenting with stroke.

Cortisol levels are routinely determined from blood, salivary or urinary samples. However, these methods do not provide information on long term cortisol secretion, accounting for the variability of HPA axis activity. There is a growing pool of evidence that shows that Hair Cortisol Concentration (HCC) examination provides a reliable retrospective estimation of integrated cortisol secretion over a period of several months. Hair grows at a rate of about 1 cm/month, thus 3 cm of hair would give an indication of the cortisol levels over the previous 3 months. HCC has been evaluated in several clinical settings in which activity of the HPA axis and cortisol levels over a period of time are of interest. Studies have demonstrated increased levels of hair cortisol in chronic stress, as well as conditions associated with stress such as pregnancy , unemployment , PTSD, alcohol withdrawal and chronic pain and more importantly, in patients admitted to hospital with acute myocardial infarction. Nevertheless, the association between hair cortisol levels and the risk for stroke has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Age of 18 years or older.

Exclusion Criteria:

* Female sex.
* Patients for whom a hair sample of at least 3cm from vertex posterior cannot be obtained.
* Hemorrhagic stroke.
* Documented atrial fibrillation or flutter during admission or at any time in the past.
* Use of inhaled, systemic or topical corticosteroids at study initiation, or during the previous 12 months.
* Disorders associated with disruption of HPA axis (Cushing syndrome, Addison syndrome).
* Bleaching or use of artificial hair color.
* Inability to sign informed consent.
* Morbid obesity (BMI > 35).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases - Consenting patients admitted to internal medicine wards with acute ischemic (non cardioembolic) stroke.
  Controls - Consenting patients admitted to internal medicine wards due to indications other than stoke or acute myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Concentration of hair cortisol | Hospital stay, on average - 24 hours from admission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Eilon Krashin, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Stalder T, Kirschbaum C. Analysis of cortisol in hair--state of the art and future directions. Brain Behav Immun. 2012 Oct;26(7):1019-29. doi: 10.1016/j.bbi.2012.02.002. Epub 2012 Feb 15. PMID 22366690